CLINICAL TRIAL: NCT03354260
Title: Personalized Adapted Diet and Nutritional Follow-up With Therapeutic Education in Critically Ill Patients : Impact on Calorie and Protein Deficit, on Weight, Mortality, and Quality of Life
Brief Title: Optimization of Oral Diet in Critically Ill Patients
Acronym: NAP-REA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of patient intube more than 5 days
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9661; 15715B-31 (Other: ANSM)
Record Dates: First submitted 2017-10-20; First posted 2017-11-27 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2017-10

CONDITIONS: Food Intake; Critically Ill Patients; Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Optimized personalized oral nutrition in ICU and nutritional follow up with therapeutic educational after exit of ICU
  Interventions: Other: Personalized adapted oral diet and nutritional education
- Control (No Intervention)

INTERVENTIONS:
Other: Personalized adapted oral diet and nutritional education — Optimized personalized oral nutrition in ICU and nutritional follow up with therapeutic educational after exit of ICU
  Arms: intervention

SUMMARY:
The purpose of the present study is to evaluate the effects of a personalized oral diet in the critically ill patients during ICU stay and after as compared usual oral diet.

DETAILED DESCRIPTION:
This is a prospective randomized controlled single center clinical trial. This trial include patient over 18 year hospitalized in ICU and ventilated more than 5 days and/or with denutrition after 5 days of no food intake in ICU without shock and/or respiratory distress. The randomization is awebsite randomization with stratification on age, presence of sepsis at inclusion, renal failure The day of the resumption of the oral feeding (J0), realization of a protocolized swallowing test then randomization and creation of a control and intervention group

Control group:

* Nutrition in resuscitation according to medical prescription: food recovery with a light meal consisting of soup and desserts and evolution to a normal meal according to the capabilities of patients
* Daily quantification of ingesta (calories and proteins) by a dietitian until the exit resuscitation. Comparison with caloric-protein targets.
* Nutritional evaluation before the release of resuscitation.

Intervention group:

* NAP: "Customized Adapted Nutrition"
* Daily quantification of ingesta (calories and proteins) by a dietitian until the exit resuscitation. Comparison with caloric-protein targets.
* Therapeutic education.
* Nutritional evaluation before the release of resuscitation.
* Creation at the exit of resuscitation of a nutritional linkage sheet with instructions food

The prospects for optimizing oral replenishment are multiple:

* reduce morbidity and mortality within 3 months after a stay in intensive care unit.
* improve autonomy and quality of life after a stay in intensive care.
* improve the privileged relationship with the patients' families.
* strengthen links within the resuscitation team and with downstream services.
* Educate patients on a nutritional level.

ELIGIBILITY:
Inclusion Criteria:

- patient 18 yo or above hospitalized in ICU and ventilated more than 5 days and/or with severe denutrition after 5 days of no food intake in ICU without shock and/or respiratory distress

Exclusion Criteria:

* age under 18 yo, pregnancy,
* protected patients
* moribund patient (life expectancy of 48h or below),
* patient with disorders of swallowing
* tracheostomy
* patient with shock and/or respiratory distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Impact on the weight 3 months after the renewal of oral intakes | at 90 days
  Decrease of weight variation 3 months after the renewal of oral intakes

SECONDARY OUTCOMES:
weight at D30 | at 30 days
  weight on the 30th day after renewal of oral intakes
mortality at D30 | at 30 days
  mortality on the 30th day after renewal of oral intakes
mortality at D90 | at 90 days
  mortality on the 90th day after renewal of oral intakes
length of stay in Intensive car unit | until the 90th day
  number of days in Intensive car unit in 3 months after renewal of oral intakes
length of stay in Hospital | until the 90th day
  number of days in Hospital in 3 months after renewal of oral intakes
length of stay in rehabilitation center | until the 90th day
  number of days in rehabilitation center in 3 months after renewal of oral intakes
infectious and non infectious complications | until the 90th day
  number and type of complication in 3 months after renewal of oral intakes
quality of life and autonomy | at 15 days
  score of autonomy Katz Score from 0 to 6
quality of life and autonomy | at 15 days
  SF 36 Score from 0 to 100
quality of life and autonomy | at 30 days
  score of autonomy Katz Score from 0 to 6
quality of life and autonomy | at 30 days
  SF 36 Score from 0 to 100
quality of life and autonomy | at 60 days
  score of autonomy Katz Score from 0 to 6
quality of life and autonomy | at 60 days
  SF 36 Score from 0 to 100
quality of life and autonomy | at 90 days
  score of autonomy Katz Score from 0 to 6
quality of life and autonomy | at 90 days
  SF 36 Score from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Celine Dupy-Richard, dietitian, Principal Investigator — Montpellier University Hospital
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided